CLINICAL TRIAL: NCT03775031
Title: Impact of Chemical Peels and Fractional Laser on IGF-1 Levels in Skin
Brief Title: Chemical Peels and Fractional Laser on IGF-1 Levels in Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Molly A. Wanner, MD, Dermatologist, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018P001770
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Chemexfoliation

STUDY DESIGN:
Intervention Model Description: Randomized-Controlled (Subjects will serve as their own control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fraxel 1927nm (Active Comparator): Treatment setting for Fraxel 1927 nm: 20 mJ, Treatment level 8, 6 passes
  Interventions: Device: Fractional Laser and Chemical Peel
- Fraxel 1550nm (Active Comparator): Treatment setting for Fraxel 1550 nm: 70 mJ, Treatment level 6, 6 passes
  Interventions: Device: Fractional Laser and Chemical Peel
- 25% TCA Peel (Active Comparator): 25% TCA on 5 x 5 cm of sun exposed back
  Interventions: Device: Fractional Laser and Chemical Peel
- Control (Placebo Comparator): Patient serves as their own control
  Interventions: Device: Fractional Laser and Chemical Peel

INTERVENTIONS:
Device: Fractional Laser and Chemical Peel — Fractional 1927 nm Laser, Fractional 1550 nm Laser, and 25% TCA (trichloroacetic acid) peel

SUMMARY:
The purpose of this study is to evaluate the impact of fractional laser versus chemical peels on IGF-1 levels in skin.

DETAILED DESCRIPTION:
This study is designed to assess the feasibility of using a fractional non ablative laser and chemical peels to wound skin, and thereby elicit a change in IGF-1. Our hypothesis is that fractional non ablative laser and a TCA chemical peel can induce similar effects as the fractional ablative laser at three months. In other words, our theory is that these approaches can stimulate the production of IGF-1 in older skin and restore UV damage repair and response mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects >55 years old
* Fitzpatrick type I-II
* Able to provide informed consent.
* Cutaneous photodamage of 3 or above on the Larnier photodamage scale (see Appendix).

Exclusion Criteria:

* Prior laser or peel treatment in the area evaluated in the current study in the past year.
* Currently taking immunosuppressant medications known to interfere wound healing or anti-inflammatory medications (such as NSAIDs, or steroids).
* Subjects who have underlying diseases that could alter wound healing response (such as Diabetes).
* Currently taking insulin.
* History of substance abuse, mental dysfunction, or other factors limiting ability to cooperate with study.
* History of abnormal scarring such as Keloids.
* History of vitiligo.
* Allergy or sensitivity or allergy to topical anesthesia
* Inability to use sunscreen.
* History of smoking in the last 10 years
* Scar or prior surgery in the area of treatment.
* Use of isotretinoin in the prior 6 months
* Subjects who have bleeding disorders or who are taking anticoagulants

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
IGF-1 Levels | 3 months
  To quantify IGF-1 levels in skin

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Clinical Unit for Research Trials and Outcomes in Skin, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No